CLINICAL TRIAL: NCT03269916
Title: Fertility and Ovarian Reserve Function in the Patient With Inflammatory Bowel - a Cross-sectional Survey and Case Control Study
Brief Title: Fertility and Ovarian Reserve Function in the Patient With Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, pengxiang, Attending doctor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SixthSunYetSen
Record Dates: First submitted 2017-08-13; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Fertility Disorders; Ovarian Reserve Function; Pregnancy Outcomes
MeSH Terms: interventions — Estrogens; Follicle Stimulating Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBD patients (Experimental): IBD patients, 17-40 years old, female
  Interventions: Other: Anti Mueller hormone; Other: Estrogen; Other: Follicle-Stimulating Hormone; Other: Antral alveolar cell count
- healthy control (Other): 17-40 years old , female, without any gynecological disease
  Interventions: Other: Anti Mueller hormone; Other: Estrogen; Other: Follicle-Stimulating Hormone; Other: Antral alveolar cell count

INTERVENTIONS:
Other: Anti Mueller hormone — used to assess ovarian reserve parameters
Other: Estrogen — used to assess ovarian reserve parameters
Other: Follicle-Stimulating Hormone — used to assess ovarian reserve parameters
Other: Antral alveolar cell count — used to assess ovarian reserve parameters

SUMMARY:
ECCO consensus, the fertility would decline in activity inflammatory bowel disease(IBD), because of anus lesions and pelvic abscess, or who underwent surgery, especially in patients with ileal pouch anal anastomosis (IPAA) storage.The study on fertility in inflammatory bowel disease were almost epidemiological investigation, the lack of objective evaluation of fertility, and controversial.This study will explore the fertility, ovarian reserve function and the pregnancy outcomes in patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

1. Inflammatory bowel disease
2. 17-40 years old
3. female

Exclusion Criteria:

1. in pregnancy or lactation
2. a drug that has been or is being used known to affect ovarian function, such as cyclophosphamide
3. reproductive system diseases unrelated to disease or treatment of inflammatory bowel disease, such as hysterectomy, pelvic radiotherapy after surgery, after ovariectomy, polycystic ovary syndrome, endometriosis, ovarian granulosa cell tumor
4. other endocrine diseases, such as prolactin, hyperthyroidism, lead to endocrine disorders;
5. malignant tumor

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
The AMH of IBD patients is lower than that of healthy women | 1 month
  AMH is used to assess ovarian reserve function
The E2 of IBD patients is lower than that of healthy women | 1 month
  E2 is used to assess ovarian reserve function
The FSH of IBD patients is lower than that of healthy women | 1 month
  FSH is used to assess ovarian reserve function
The AFC of IBD patients is lower than that of healthy women | 1 month
  AFC is used to assess ovarian reserve function

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhi, PHD, Study Chair — The Sixth Affiliated Hospital of Zhongshan University
Locations (1):
- The Sixth Affiliated Hospital of Zhongshan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided